CLINICAL TRIAL: NCT05219656
Title: Long-term Outcome of Patients With Acute Ulcerative Colitis Treated With Cyclosporine Rescue Therapy.
Brief Title: Efficacy of Cyclosporine Rescue Therapy in Acute Ulcerative Colitis.
Acronym: Cyclo
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Heli T Eronen, MD, Kanta-Häme Central Hospital
Other Study IDs: R19617
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Ulcerative Colitis Acute
Keywords: Cyclosporine A; Rescue therapy
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cyclosporine A — Rescue therapy in acute severe ulcerative colitis
  Other Names: CyA

SUMMARY:
The efficacy and safety of Cyclosporine A as rescue therapy for acute severe ulcerative colitis in long-term follow-up.

DETAILED DESCRIPTION:
All UC patients treated with CyA in Tampere University Hospital between 2009 and 2018 were reviewed from patient records and analyzed. Amelioration of UC was defined as clinical response for rescue therapy with no need for colectomy or third-line rescue therapy at the same hospitalization as index flare. Relapse was defined as requiring further Cs treatment, re-hospitalization, biologicals, small molecules, or colectomy later in follow-up. Patients were followed-up from the date of index flare until colectomy, death, or the end of observation period. Adverse events related to treatment were assessed throughout the duration of treatment. Surgical complications were defined by using Clavien-Dindo classification (grade III-V classified as severe complications). The surgical complications in Cyclosporine-treated patients were compared to all patients operated for treatment refractor UC in Tampere University Hospital within the same follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to hospital for acute flare of UC and treated with CyA rescue therapy.
* Age 16 or over

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated in Tampere University Hospital with Cyclosporine rescue therapy for acute flare of UC.
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Response | From january 2009 to december 2018
  Clinical response for CyA with no need for colectomy or further enhancement of treatment with infliximab at the same hospitalization ad index flare
Remission | From january 2009 to december 2018
  Remission was defined as no need for further corticosteroids, re-hospitalization, enhancement of treatment with biologicals or small molecules or colectomy within follow-up.
Adverse events | From january 2009 to december 2018
  Reported treatment related adverse events.
Surgical complications | From January 2009 to December 2018
  Reported surgical complications.

CONTACTS AND LOCATIONS:
Overall Officials: Heli Eronen, Principal Investigator — Kanta-Häme Central Hospital

IPD SHARING:
Plan to Share IPD: No